CLINICAL TRIAL: NCT00699894
Title: Comparison of Aprepitant PO and Ondansetron IV for Prevention of Postoperative Nausea and Vomiting (PONV) in Patients Undergoing Orthognathic Surgery and General Anesthesia.
Brief Title: Aprepitant PO vs Ondansetron IV for Prevention of Postoperative Nausea and Vomiting
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistical difficulties running the study
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 07118
Record Dates: First submitted 2008-06-16; First posted 2008-06-18 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-08

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: PONV; prevention of postoperative nausea and vomiting; aprepitant; ondansetron; orthognathic surgery
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Vomiting | interventions — Aprepitant; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): aprepitant 40 mg + normal saline IV
  Interventions: Drug: aprepitant 40 mg
- 2 (Active Comparator): placebo PO + ondansetron 4 mg IV
  Interventions: Drug: ondansetron 4 mg

INTERVENTIONS:
Drug: aprepitant 40 mg — aprepitant 40 mg PO 1-3 hours prior to surgery
  Other Names: emend 40 mg
  Arms: 1
Drug: ondansetron 4 mg — ondansetron 4 mg IV 2-5 minutes prior to induction of anesthesia
  Other Names: zofran 4 mg
  Arms: 2

SUMMARY:
Postoperative nausea and vomiting (PONV) persists as one of the more common complications of surgery. Although rarely life-threatening, it is the postoperative outcome that is most unfavorable to patients, even more undesirable than pain. Orthognathic surgery corrects conditions of the jaws and face related to structure, growth, sleep apnea, bad bite, or congenital malformations. The bones of the face and jaws are cut and placed in a new position. There is a high rate of PONV in orthognathic surgery (56%). It is particularly challenging to the patient as their jaws are kept closed together with wires or elastic bands. Nausea in a patient with restricted mouth opening can be psychologically unnerving and puts them at risk for fluid in their lungs.

Gan and colleagues showed a higher efficacy of aprepitant over ondansetron in preventing PONV and nausea severity after open abdominal surgery. From this study, the FDA approved the use of aprepitant for PONV prevention in patients >18 years of age. Gan suggested further investigation in different populations.

Our randomized, double-blind, prospective study will compare the efficacy of aprepitant PO versus ondansetron IV in a high risk setting for PONV: adolescents undergoing orthognathic surgery.

Our study will involve 200 consecutive, adolescent patients (ages 15-25) who will undergo at least a Le Fort 1 osteotomy (upper jaw surgery) under general anesthesia and require hospital admission for at least one night. We will exclude patients who are currently taking medications that have interactions with aprepitant (pimozide, terfenadine, astemizole, cisapride), those who have a known vomiting disorder such as bulimia, and those who have vomited for any reason within 24 hours of surgery. The procedure will be performed by 5 surgeons and general anesthesia will be administered by 3 anesthesiologists at one institution. A study coordinator, who will not be involved in the treatment, will create the randomization schedule in order to ensure blindness. The patients will be randomized to either of two groups: 1) aprepitant 40 mg PO 2) ondansetron 4 mg IV. Appropriate verbal and written consent will be obtained by the priniciple investigator or surgeon.

On the day of the procedure, all patients will receive a pill (aprepitant or aprepitant placebo) at least 1 hour prior to induction of anesthesia and an IV infusion (ondansetron or saline) over 2-5 minutes prior to intubation. The timing and doses of medications will be consistent with manufacturer's recommendations. An established protocol will ensure every patient will receive the same anesthetic regiment. Patient's fluid status will be closely monitored and hydrated appropriately according to known fluid balance calculations.

Efficacy will be assessed based on criteria set by Gan et al and will be based on the presence/absence of a vomiting episode, use of rescue medication and subjective evaluation of nausea. Patients will be monitored continuously in the PACU and on the hospital floor by the caring team (nurse, resident, anesthesiologist, surgeon) for any emetic episode or use of rescue therapy. An emetic episode is defined as an act of vomiting (oral expulsion of stomach contents) or retching (non-productive vomiting). Nausea will be assessed at intervals of 0, 2, 6, 24 hours after surgery with T0 being time of extubation. Patients will rate nausea on a 11-point verbal rating scale, with 0 being "not nausea" to 10 being "the worst nausea." Rescue medication will be offered if the patient has more than one episode of vomiting or retching, if the patient has nausea lasting longer than 15 minutes, or if the patient requests it for established nausea or vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 15-25 who have reached skeletal maturity and are scheduled for Le Fort 1 osteotomy as part of standard care.
* Capable of providing informed consent.

Exclusion Criteria:

* Patients with hypersensitivity to medications contraindicated with aprepitant: pimozide, terfenadine, astemizole, cisapride.
* Patients with a known vomiting disorder
* Patients who have vomited for any reason within 24 hours prior to surgery.
* Patients who are pregnant or nursing.
* Patients who are unable to provide informed consent.

Ages: 15 Years to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2008-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
No vomiting and use of rescue medications | 24 hours

SECONDARY OUTCOMES:
no nausea based on verbal rating scale | 0, 2, 6, 24 hours
time to first emetic episode | 24 hours
time to use of rescue medications | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Choi, DDS, Principal Investigator — Long Island Jewish Medical Center
Locations (1):
- Long Island Jewish Medical Center/Schneider's Children Hospital, New Hyde Park, New York, United States

REFERENCES:
- [Background] Gan TJ, Apfel CC, Kovac A, Philip BK, Singla N, Minkowitz H, Habib AS, Knighton J, Carides AD, Zhang H, Horgan KJ, Evans JK, Lawson FC; Aprepitant-PONV Study Group. A randomized, double-blind comparison of the NK1 antagonist, aprepitant, versus ondansetron for the prevention of postoperative nausea and vomiting. Anesth Analg. 2007 May;104(5):1082-9, tables of contents. doi: 10.1213/01.ane.0000263277.35140.a3. PMID 17456656